CLINICAL TRIAL: NCT02105545
Title: Genome Sequencing of Human Cancer Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INST 1306
Record Dates: First submitted 2014-03-13; First posted 2014-04-07 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: cancer; oncology; malignant; malignancy; genetics; genomics; exome; DNA; RNA; sequencing; epigenetic; clinically actionable findings; CAF; secondary findings; SF; single nucleotide variants; SNV; bioinformatics; genotype; The American College of Medical Genetics and Genomics; ACMG
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cancer Treatment Options (Experimental): Blood samples and, for some patients, buccal (mouth cell) samples will be collected at diagnosis and/or relapse. Solid tumor samples will be collected in the normal course of treatment, from biopsy, blood or other specimens. For blood-based cancers such as leukemia, blood and bone marrow specimens will be collected before treatment begins, on day 29 and possibly at a later time point if relapse occurs.
  Interventions: Other: Cancer Treatment Options

INTERVENTIONS:
Other: Cancer Treatment Options — Patients may meet, depending on test results, with their physician and a genetic counselor to discuss possible changes in their treatment options and/or lifestyle changes.
  Other Names: treatment options; lifestyle changes; behavioral changes; genetics

SUMMARY:
The goal of this study is to develop a new, local system that will use special tests based on patients' genetic makeup to better tailor cancer care at the University of New Mexico Cancer Center.

The Food and Drug Administration has already approved over forty (40) drugs to treat cancer patients based on specific genetic makeup, and more agents are in development that will support this new approach to treatment, often referred to as "personalized medicine."

The goal of performing specific tests on patients' genetic material is to discover tumor-specific, single nucleotide variations (SNVs) and other forms of genetic changes (called epigenetic changes) that can be detected when comparing normal tissue and tumor tissue. This can help guide cancer care decisions that may be more effective for patients. These will be called clinically actionable findings, or CAF.

Additional health related findings may be made, not related to cancer but to other conditions, diseases or syndromes. These are called secondary findings (SF). In this study the investigators will also measure how often they find SF and will discuss their possible impact on other aspects of patients' health. If patients want to know about these findings, they will be discussed with a panel of experts including genetic counselors.

Finally, the investigators will compare how often CAF and SF differ from those identified in nationwide samples.

DETAILED DESCRIPTION:
For brevity, the investigators include the approaches of whole genome sequencing, whole exome sequencing of just the protein-coding exons, enrichment and sequencing of methylated DNA and RNA or transcriptome-sequencing under the broad category term, Whole Genome Sequencing (WGS).

The development of rapid and low cost next-generation genome sequencing technologies brings the promise of a new era of precision therapeutics to clinical practice, but it is associated with significant challenges, including reproducible generation of high-quality sequence data and the need for comprehensive data analysis and interpretation that is translatable to clinical action. Equally critical are the ethical, legal, and social issues surrounding the introduction of WGS testing and its clinical application in multiethnic, multicultural populations, particularly those who have historically experienced discrimination or even unethical research practices. Of particular concern are issues surrounding the privacy, ownership, storage, and use of WGS data.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a malignant diagnosis at the time of diagnosis or relapse
* Any age (minimum 0 days old)
* Male or Female
* Pregnant women are eligible for this study
* Patients may have existing, non-oncological genetic disorders
* Patients may have received any amount of prior treatment
* Participants (or their parent/legal guardian in the case of minors) must have the ability to understand and the willingness to sign a written informed consent or assent form

Exclusion Criteria:

* Subjects for whom sufficient cancer tissues are not available to meet the objectives of the study.
* Cognitively impaired adults are excluded from participation
* Adults not able to consent for themselves are excluded from participation
* Prisoners may not participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically actionable findings | 3 years
  The investigators will utilize new genomics technologies in to identify potentially Clinically Actionable Findings (CAF) in patient tumor and other samples. Based on individual patient data, alternative treatment options will be offered to patients.

SECONDARY OUTCOMES:
Frequency of findings (CAF) in cancer patients treated locally | 3 years
  The investigators will measure the frequency with which clinically actionable findings (CAF) that could impact current patient care decisions occur in tumor and other samples.
Percentages and types of local patient CAF aligned with national genomics data sets | 3 years
  Determine whether CAF identified in the unique patient populations treated at the University of New Mexico Cancer Center differ from those identified in nationwide data sets such as The 1000 Genomes Project or The Cancer Genome Atlas (TCGA) data collections.
Number of barriers limiting use of genomics information in local patient care | 3 years
  Identify the numbers and types technological, social, ethical and/or legal barriers that might limit the use of genomics information in patient care at the University of New Mexico Cancer Center and the University of New Mexico Health Sciences Center. The investigators will assess the frequency of use of CAF by local treating physicians. They will assess how often cancer treatment choice is altered as a result of providing CAF to physicians and patients. The investigators will assess how often identified CAF are entered into patient medical records. They will assess the frequency with which patients choose to receive information about potentially detrimental SF unrelated to their cancer care.
Percentage of patients with secondary findings (SF) | 2 years
  Identify other genomics-based findings in patient samples unrelated to cancer care, but which might impact other aspects of patients' health. These will be referred to as Secondary Findings, or SF. For example, if a SF is identified that suggests an increased risk of diabetes, this would be considered a secondary finding. This will be discussed by a panel of medical experts, and if patients wish to have this information returned to them, their doctor and genetic counselor will discuss the SF. Patients can choose not to have SF returned to them.
Percentages and types of local patient Secondary Findings aligned with national genomics data sets | 3 years
  Determine whether SF identified in the unique patient populations treated at the University of New Mexico Cancer Center differ from those identified in nationwide samples such as The 1000 Genomes Project or The Cancer Genome Atlas (TCGA).

CONTACTS AND LOCATIONS:
Overall Officials: Stuart S Winter, MD, Study Chair — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org